CLINICAL TRIAL: NCT03363750
Title: Pilot Study of Mind-Body Skills Groups for Adolescents With Depression in Primary Care
Brief Title: Study of Mind-Body Skills Groups for Adolescents With Depression in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: The Center for Mind-Body Medicine (Other); Eskenazi Health (Other)
Responsible Party: Principal Investigator, Michelle Salyers, Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1707293729
Record Dates: First submitted 2017-11-21; First posted 2017-12-06 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Depression; Depressive Disorder
Keywords: Depression; Adolescent; mind-body-skills; group therapy; primary care
MeSH Terms: conditions — Depression; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mind-body-skills intervention (Experimental): mind-body-skills group intervention offered weekly for 10 weeks
  Interventions: Behavioral: mind-body-skills group

INTERVENTIONS:
Behavioral: mind-body-skills group — mind-body skills group program incorporates meditation, guided imagery, breathing techniques, autogenic training, biofeedback, genograms, and self-expression through words, drawings, and movement

SUMMARY:
The Center for Mind -Body Medicine has developed a mind-body skills group program that incorporates meditation, guided imagery, breathing techniques, autogenic training, biofeedback, genograms, and self-expression through words, drawings, and movement. These mind-body skills are designed to increase self-awareness and self-regulation. This program has been shown to significantly improve depression symptoms in children and adolescents with posttraumatic stress disorder in Gaza, but it has not yet been tested in a US adolescent population. The purpose of this study is to determine the feasibility of using mind-body skills groups to reduce depression in adolescents and to investigate the effects of the program on factors such as self-efficacy, mindfulness and rumination which are likely to mediate improvement.

ELIGIBILITY:
Inclusion Criteria:

* Eskenazi Primary Care patients at time of screening
* 13-17 years old
* Diagnosis of depression confirmed by Mini International Neuropsychiatric Interview (MINI) Kid Screen (with adolescent)
* English speaking
* Willingness to attend mind body skills group for duration of the intervention (10 sessions over approximately 10 weeks)

Exclusion Criteria:

* History of bipolar disorder or psychosis
* Acute and immediate risk of suicide, determined by clinical assessment
* Lack of capacity to assent (adolescent) or lack of capacity to consent (parent/guardian)
* Previous participation by the adolescent in the Eskenazi Mind Body Group intervention

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
Change in Children's Depression Inventory-2 (CDI-2) scores | from baseline to within one month after end of intervention
  self report long version (28 items) to assess the presence and severity of depressive symptoms in children
Change in Children's Depression Inventory-2 (CDI-2) scores | from baseline to approximately 3 months after end of intervention
  self report long version (28 items) to assess the presence and severity of depressive symptoms in children

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) score | from baseline to within one month after end of intervention
  self report (9 questions) to screen for the presence and severity of depression
Change in Patient Health Questionnaire-9 (PHQ-9) score | from baseline to approximately 3 months after end of intervention
  self report (9 questions) to screen for the presence and severity of depression
Change in Rumination Subscale of the Children's Response Style Questionnaire Score | from baseline to within one month after end of intervention
  self report (13 questions) of rumination symptoms
Change in Rumination Subscale of the Children's Response Style Questionnaire Score | from baseline to approximately 3 months after end of intervention
  self report (13 questions) of rumination symptoms
Change in Mindful Attention Awareness Scale-Adolescent (MAAS) score | from baseline to within one month after end of intervention
  self report (14 questions) designed to assess open or receptive awareness of and attention to what is taking place in the present
Change in Mindful Attention Awareness Scale-Adolescent (MAAS) score | from baseline to approximately 3 months after end of intervention
  self report (14 questions) designed to assess open or receptive awareness of and attention to what is taking place in the present
Change in Self-Efficacy Questionnaire for Depression in Adolescents (SEQ-DA) score | from baseline to within one month after end of intervention
  self report (12 items) designed to measure self-perceived ability to cope with depressive symptoms
Change in Self-Efficacy Questionnaire for Depression in Adolescents (SEQ-DA) score | from baseline to approximately 3 months after end of intervention
  self report (12 items) designed to measure self-perceived ability to cope with depressive symptoms
Change in Suicide Ideation Questionnaire (SIQ) score | from baseline to within one month after end of intervention
  self report (30 or 15 items depending on grade level) to assess frequency of suicidal ideation
Change in Suicide Ideation Questionnaire (SIQ) score | from baseline to approximately 3 months after end of intervention
  self report (30 or 15 items depending on grade level) to assess frequency of suicidal ideation
Acceptability Questionnaire | within one month after end of intervention
  self report (15 items) intervention acceptability assessment of usefulness and helpfulness of the intervention
Acceptability Questionnaire | approximately 3 months after end of intervention
  self report (15 items) intervention acceptability assessment of usefulness and helpfulness of the intervention
Acceptability Questionnaire - open-ended questions for qualitative analyses | within one month after end of intervention
  3 open-ended questions to gather qualitative data about the usefulness and helpfulness of the intervention
Acceptability Questionnaire - open-ended questions for qualitative analyses | approximately 3 months after end of intervention
  3 open-ended questions to gather qualitative data about the usefulness and helpfulness of the intervention
Change in Hope Scale Score | from baseline to within one month after end of intervention
  * self report (12 items), 4-point Likert scale(1=Definitely False to 4=Definitely True)
  * evaluates global hope (range 8-32); there are also 2 subscales: hope agency (range 4-16) and hope pathways (range 4-16)
  * includes distracter items
  * global hope score calculated by summing the hope agency and hope pathways scores (omitting distracter items)
  * higher scores indicate a person has higher hope
Change in Hope Scale Score | from baseline to approximately 3 months after end of intervention
  * self report (12 items), 4-point Likert scale(1=Definitely False to 4=Definitely True)
  * evaluates global hope (range 8-32); there are also 2 subscales: hope agency (range 4-16) and hope pathways (range 4-16)
  * includes distracter items
  * global hope score calculated by summing the hope agency and hope pathways scores (omitting distracter items)
  * higher scores indicate a person has higher hope
Change in Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) Score | from baseline to within one month after end of intervention
  * self report (14 items) to measure positive affect, satisfying interpersonal relationships, and positive functioning
  * 5-point Likert scale (1=none of the time to 5=all of the time)
  * total score is calculated by summing each item score (range 14-70)
  * higher scores represent increased levels of mental wellbeing
Change in Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) Score | from baseline to approximately 3 months after end of intervention
  * self report (14 items) to measure positive affect, satisfying interpersonal relationships, and positive functioning (range 14-70)
  * 5-point Likert scale (1=none of the time to 5=all of the time)
  * total score is calculated by summing each item score (range 14-70)
  * higher scores represent increased levels of mental wellbeing

CONTACTS AND LOCATIONS:
Overall Officials: Michelle P Salyers, PhD, Principal Investigator — Indiana University
Locations (1):
- Eskenazi Health Primary Care, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cunningham LD, Salgado EF, Aalsma MC, Garabrant JM, Staples JK, Gordon JS, Salyers MP. Do adolescents consider mind-body skills groups an acceptable treatment for depression: results from a pilot study. BMC Pediatr. 2021 Oct 27;21(1):475. doi: 10.1186/s12887-021-02942-3. PMID 34706710